CLINICAL TRIAL: NCT07050069
Title: The Effect of Threshold Pressure-loaded Respiratory Muscle Training Combined With Transcranial Intermittent Theta Burst Stimulation on Respiratory Function in Patients With Spinal Cord Injury
Brief Title: Effect of Threshold Pressure-Loaded RMT + tTBS on Respiratory Function in SCI Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Xue Jiang, Associate Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024PS1936K
Record Dates: First submitted 2025-06-16; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Group A: sham stimulation + threshold pressure-loaded respiratory muscle training; Group B: iTBS + traditional respiratory training; Group C: iTBS + threshold pressure-loaded respiratory muscle training.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: sham stimulation + threshold pressure-loaded respiratory muscle training (Experimental): Sham Stimulation "8" coil at bilateral diaphragmatic cortical projections (2-3 cm ant. to coronal line, 3 cm lat. to midline). 80% MT intensity. Each pulse train: 3 bursts (50 Hz intra/5 Hz inter), 2s on/8s off. Total 1,200 pulses (600/side), 5 sess/wk × 20 sess. Coil at 90° to scalp to avoid cortical current.
  Threshold Pressure-Loaded RMT Saike trainer used. Pt. seated/reclined, nasal clips occluding nares. Filter mouthpiece connected to valve; tight oral seal. Resistance: 30% of MIP/MEP. 10 min inhale/exhale each, 20 min/d. Weekly MIP/MEP reassessment to adjust resistance. 4 wk, 5 d/wk.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) Device / Respiratory Training Device
- Group B: iTBS + traditional respiratory training (Experimental): iTBS Therapy 8-shape coil at bilateral diaphragmatic cortical projections (2-3 cm ant. to coronal line, 3 cm lat. to midline). 80% MT. Each pulse train: 3 bursts (50 Hz intra/5 Hz inter), 2s on/8s off. Total 1,200 pulses (600/side), 5 sess/wk × 20 sess.
  Traditional Respiratory Training 5 therapist-led maneuvers: Pursed-lip: inhale (3-4s) via nose, pause (1-2s), exhale (5-6s) with pursed lips (6-8 br/min), 20 br/set.
  Diaphragmatic: seated/supine, hands over umbilicus. Inhale to expand abdomen (3-5s), exhale to compress (6-8s). 4-6 br/min, 20 br/set.
  Forced exhale: inhale (3-5s), forcefully exhale "ha" (2-3s), 4-6 br/min, 20 br/set.
  Resisted inhale: supine, 1kg sandbag on umbilicus. Diaphragmatic breathing (4-6 br/min), 20 br/set.
  3 sets/d, 5d/wk × 4wk.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) Device / Respiratory Training Device
- Group C: iTBS + threshold pressure-loaded respiratory muscle training (Experimental): iTBS Therapy 8-shape coil at bilateral diaphragmatic cortical projections (2-3 cm ant. to coronal line, 3 cm lat. to midline). 80% MT. Each pulse train: 3 bursts (50 Hz intra/5 Hz inter), 2s on/8s off. Total 1,200 pulses (600/side), 5 sess/wk × 20 sess.
  Threshold Pressure-Loaded RMT Saike trainer used. Pt. seated/reclined, nasal clips occluding nares. Filter mouthpiece connected to valve; tight oral seal. Resistance: 30% of MIP/MEP. 10 min inhale/exhale each, 20 min/d. Weekly MIP/MEP reassessment to adjust resistance. 4 wk, 5 d/wk.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS) Device / Respiratory Training Device

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) Device / Respiratory Training Device — Participants received group-specific interventions 5 days/week for 4 weeks.

SUMMARY:
The purpose of this clinical trial is to understand whether threshold pressure load respiratory muscle training combined with iTBS can effectively improve the respiratory function of SCI patients. The main questions it aims to answer are:

* The impact of threshold pressure load respiratory muscle training on the respiratory function of SCI patients.
* The impact of iTBS treatment at the cortical projection point of the diaphragm on the respiratory function of SCI patients.
* Whether the combination of the above two treatment techniques is superior to single treatment.

DETAILED DESCRIPTION:
Researchers will combine threshold pressure load respiratory muscle training and transcranial iTBS and compare them with single treatments to see if the combined treatment is superior to single treatment.

Participants will:

* Undergo threshold pressure load respiratory muscle training or transcranial iTBS treatment or a combination of both daily for 4 weeks.
* Visit the hospital for check-ups and tests every 2 weeks.
* Record their symptoms and respiratory function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spinal cord injury (SCI) meeting the 2019 revised International Standards for Neurological Classification of Spinal Cord Injury by the American Spinal Injury Association (ASIA), confirmed by CT/MRI.
* Aged 18-80 years.
* Time since injury: 2 weeks to 6 months, with spinal shock resolved.
* Injury level at T12 or above, ASIA Impairment Scale (AIS) grade A-C.
* Patients providing written informed consent after study explanation.

Exclusion Criteria:

* Patients with severe cardiorespiratory diseases (e.g., pneumothorax).
* Unstable vital signs (e.g., hypotension, arrhythmia).
* Cognitive/psychiatric disorders precluding cooperation.
* Requiring mechanical ventilation.
* Congenital spinal/limb deformities.
* Contraindications to magnetic stimulation: intracranial metal implants, pacemakers, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure | Week 0 , Week 2 , Week 4
  the maximum negative pressure generated in the respiratory system during a maximal inhalation against a closed airway, measured in cmH₂O to assess inspiratory muscle strength.
Maximal Expiratory Pressure | Week 0 , Week 2 , Week 4
  the maximum positive pressure generated in the respiratory system during a maximal exhalation against a closed airway, measured in cmH₂O to assess expiratory muscle strength.
Peak Expiratory Flow | Week 0 , Week 2 , Week 4
  the maximum speed of air flow during a forced exhalation, measured in liters per minute (L/min) to assess airway patency and respiratory function.
Peak Inspiratory Flow | Week 0 , Week 2 , Week 4
  the maximum speed of air flow during a forced inhalation, measured in liters per minute (L/min) to evaluate inspiratory muscle function and airway resistance during inhalation.
Forced Expiratory Volume in 1 second | Week 0 , Week 2 , Week 4
  the volume of air exhaled forcefully within the first second of a maximal expiratory effort, measured in liters to assess airway obstruction and lung function.
Forced Vital Capacity | Week 0 , Week 2 , Week 4
  the total volume of air exhaled forcefully and completely after a maximal inhalation, measured in liters to evaluate lung function and airway patency.

SECONDARY OUTCOMES:
Diaphragmatic Thickness | Week 0 , Week 2 , Week 4
  Position patient supine with arms up. Place convex probe at mid-axillary line (7th-9th intercostal space), parasagittal plane.
  Identify diaphragmatic muscle between pleural and peritoneal interfaces, 2-3 cm from central tendon.
  Measure thickness at end-expiration and end-inspiration (3 trials each). Calculate DTF to assess diaphragmatic function.
Diaphragmatic Displacement | Week 0 , Week 2 , Week 4
  Position patient supine/semi-recumbent, expose lower chest. Place convex probe at mid-axillary line (8th-10th intercostal space), sagittal plane.
  Visualize diaphragmatic-liver interface (right hemidiaphragm preferred). Use M-mode to record diaphragmatic movement over respiratory cycles. Measure vertical distance between end-expiration and end-inspiration positions (normal >1.5 cm for weaning).
Diaphragmatic Thickening Fraction | Week 0 , Week 2 , Week 4
  Measure Thickness at End-Expiration:
  Using ultrasound, measure the diaphragm thickness at the end of a quiet exhalation (when the diaphragm is relaxed).
  Measure Thickness at End-Inspiration:
  Measure the thickness at the end of a maximal inhalation (when the diaphragm is fully contracted).
  Calculate the Difference:
  Subtract the end-expiration thickness from the end-inspiration thickness.
  Normalize by End-Expiration Thickness:
  Divide the difference by the end-expiration thickness, then multiply by 100 to get a percentage.

OTHER OUTCOMES:
4th Intercostal Space Thoracic Mobility | Week 0 , Week 2 , Week 4
  At the 4th intercostal space along the midclavicular or anterior axillary line, thoracic mobility is measured by the difference in circumferences between maximal exhalation and inhalation using a non-stretch tape.
Maximum Vowel Prolongation Time | Week 0 , Week 2 , Week 4
  Maximum vowel prolongation time is obtained by measuring the duration of sustained /a:/ phonation from maximal inspiration to complete expiration, with the subject seated upright and maintaining consistent pitch and loudness
The incidence of pneumonia during hospitalization for each patient group | Week 0 , Week 2 , Week 4
  The incidence of pneumonia during hospitalization for each patient group is calculated as the number of newly diagnosed pneumonia cases divided by the total number of patients in the group, typically expressed per 100 patient-days or as a percentage.
Motor Function | Week 0 , Week 2 , Week 4
  Trunk Control Test,Modified Barthel Index
Hemodynamic Changes " BP " During Supine-to-Sitting Transfer | Week 0 , Week 2 , Week 4
  Measure baseline supine BP after 10-min rest.
Hemodynamic Changes "HR" During Supine-to-Sitting Transfer | Week 0 , Week 2 , Week 4
  Measure baseline supine HR after 10-min rest.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Xue, Principal Investigator — Rehabilitation Center of Shengjing Hospital, China Medical University
Locations (1):
- Rehabilitation Center of Shengjing Hospital, China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No